CLINICAL TRIAL: NCT05043298
Title: A Phase Ia/Ib Open-Label, Multi-Center Clinical Trial to Evaluate Safety, Tolerability, Pharmacokinetics and Preliminary Efficacy of IBI360 Monotherapy or in Combination With Sintilimab and (or) Chemotherapy in Advanced or Metastatic Solid Tumors
Brief Title: A Phase Ia/Ib Clinical Trial of IBI360 Monotherapy or in Combination With Sintilimab and (or) Chemotherapy in Advanced or Metastatic Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Innovent Biologics (Suzhou) Co. Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CIBI360A101
Record Dates: First submitted 2021-09-05; First posted 2021-09-14 (Actual); Last update posted 2024-10-17 (Actual); Status verified 2024-10

CONDITIONS: Advanced Solid Tumor
Keywords: Advanced Solid Tumor

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- IBI360 (Experimental)
  Interventions: Drug: IBI 360 Injection
- IBI 360 + Sintilimab (Experimental)
  Interventions: Drug: IBI 360 Injection Sintilimab

INTERVENTIONS:
Drug: IBI 360 Injection — IBI 360 dose level of escalation IV Q3W Day 1
  Arms: IBI360
Drug: IBI 360 Injection Sintilimab — IBI 360 dose level of escalation IV Q3W Day 1 Sintilimab 200mg IV Q3W Day 1
  Arms: IBI 360 + Sintilimab

SUMMARY:
This is an open label Phase Ia/Ib trial to evaluate safety, tolerability, pharmacokinetics and preliminary efficacy of IBI360 monotherapy in Advanced or Metastatic Solid Tumors

DETAILED DESCRIPTION:
Phase Ia is dose escalation and dose expansion study of IBI360 monotherapy and IBI360 in combination with sintilimab in advanced or metastatic Solid Tumors; Phase Ib is an multi-cohort trial of pancreatic carcinoma, HER2 negative gastric adenocarcinoma, advanced or metastatic solid tumors to evaluate safety and preliminary efSficacy of IBI360 in combination with sintilimab and (or) chemotherapy or IBI360 monotherapy.

ELIGIBILITY:
Inclusion Criteria:

1. Provide signed informed consent;
2. Male or female aged at 18-75 (inclusive) years;
3. Expected survival ≥12 weeks;
4. ECOG PS score 0 or 1;
5. Provide archival or fresh tissues for CLDN18.2 expression analysis;
6. Adequate laboratory parameters;
7. Suffer from advanced or metastatic malignant local solid tumors confirmed by histological diagnosis and meet the criteria of the enrolled group as follows:

Ia: The subjects for whom no standard treatment regimens are available or who is intolerable to standard treatments.

Ib: pancreatic carcinoma, HER2 negative gastric adenocarcinoma, advanced or metastatic solid tumors

Exclusion Criteria:

1. The subjects who received the treatment with CLDN18.2 monoclonal antibody or CLDN-18.2 CART;
2. The subjects who received other anti-tumor medication within 4 weeks prior to the initial dose of the study drug;
3. Any toxicity due to previous anti-tumor therapy that has not yet resolved to NCI CTCAE v5.0 grade 0 or 1 prior to the first dose of study treatment;
4. The subjects with history of hypersensitivity to the study drug;
5. The subjects were not recovery after surgery with history of gastrointestinal perforation or fistula within 6 months prior to the enrollment;
6. The subjects with symptomatic central nervous system (CNS) metastasis or carcinomatous meningitis;
7. The subjects with pyloric obstruction;
8. The subjects with active or poorly controlled serious infections

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2021-10-27 (Actual); Primary Completion 2023-08-30 (Actual); Study Completion 2023-08-30 (Actual)

PRIMARY OUTCOMES:
Safety and tolerance | up to 90 days following last dose
  Participant safety is characterized by frequency and severity of adverse events(according to NCI CTCAE 5.0)
Recommended Phase 2 Dose (RP2D) | up to 21 days following last dose level
  A recommended phase 2 dose will be determined based on safety data including dose limiting toxicities, preliminary efficacy data, and PK data

SECONDARY OUTCOMES:
Efficacy | Subjects were randomized 6 months and 1 year later
  Tumor response will be determined by the revised Response Evaluation Criteria in Solid Tumors version 1.1 (RECISTv1.1).
Pharmacokinetics | Up to 48 weeks following first dose
  Area under plasma concentration vs time curve(AUC)
Immunogenicity | up to 90 days following last dose
  Incidence of anti-drug antibodies (ADA) will be measured
Pharmacokinetics | Up to 48 weeks following first dose
  Peak plasma concentration(Cmax)
Pharmacokinetics | Clearance（CL）
  Up to 48 weeks following first dose
Pharmacokinetics | Up to 48 weeks following first dose
  Apparent volumeof distribution（V）
Pharmacokinetics | Up to 48 weeks following first dose
  Terminal Half Life（T1/2）

CONTACTS AND LOCATIONS:
Locations (1):
- Innovent Biologics (suzhou) Co. , Ltd., Suzhou, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No